CLINICAL TRIAL: NCT01842750
Title: The Use of Rectal Balloons in Radical Pelvic Radiotherapy - a Feasibility Study
Acronym: BRAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Julie Stratford, research radiographer, The Christie NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 11_RADIO_101
Record Dates: First submitted 2013-04-17; First posted 2013-04-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endorectal Balloon insertion (Experimental): A cone Beam scan will be performed prior to balloon insertion and then again with balloon in situ. The scans will be compared to see if the organs are stabilised. Questionnaires will be completed by the radiographer and the patient.
  Interventions: Device: Endorectal Balloon insertion

INTERVENTIONS:
Device: Endorectal Balloon insertion

SUMMARY:
This study aims to test the hypothesis that insertion of an endorectal balloon into a patient receiving radical prostate radiotherapy by treatment radiographers is feasible without the patient experiencing undue discomfort. In addition this study will test the hypotheses that insertion of the rectal balloon prior to radiotherapy delivery stabilises rectal volume during radiotherapy treatment and minimises organ motion within the pelvis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* ECOG performance status 0-2 (Patients with PS-2 as a result of comorbidity will be excluded).
* Patients with histologically confirmed diagnosis of prostate adenocarcinoma
* Patients who are going to undergo treatment with radical radiotherapy for prostate cancer.
* Patients must be able to receive and understand verbal and written information regarding the study and give written, informed consent
* Patients must be able to comply with trial requirements.

Exclusion Criteria:

* Patients must not have a history of previous bowel surgery involving the rectum or anus.
* Evidence of significant clinical disorder or laboratory finding which, in the opinion of the investigator makes it undesirable for the patient to participate in the trial, as well as any other serious uncontrolled medical condition.
* Any patient with a medical or psychiatric condition that impairs their ability to give informed consent
* Pre-existing anorectal disease, e.g. Haemorrhoids, active bleeding, anal irritation, inflammatory bowel disease.
* Patients who are unable to give consent.
* Patients in clinical trials of new investigational medicinal products or treatment regimens unless there is written, prior agreement that the patient can also consent to this study, and that clinical data can also be used for this study.
* Prior pelvic radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Tolerability | Patients will be assessed for 4 weeks throughout radiotherapy treatment
  The primary aim is to determine whether the balloon insertion is tolerated throughout treatment. The principle outcome measure is the percentage of patients who tolerate the endorectal balloon throughout treatment.

SECONDARY OUTCOMES:
rectal volume | patient scans will be reviewed over 4 weeks of radiotherapy
  Rectal volume stability will be determined by comparing the rectal volume for scans with the endorectal balloon(ERB)in situ to scans without the ERB in situ
Assessment of planning target volume (PTV) coverage | patients will be reviewed across a 4 week radiotherapy treatment period.
  PTV coverage and an assessment of prostate shape and position between the weekly imaging scans with the balloon in situ will be compared with the position of the prostate and PTV coverage on the original planning scan with the balloon in situ
Rectal wall sparing | patients reviewed across 4 weeks of radiotherapy treatment
  Rectal wall sparing will be assessed by comparing the estimated dose determined from the imaging scans with the ERB in situ and not in situ against the planned dose from the radiotherapy planning scan
Acute toxicity | patients toxicity will be assessed over 4 weeks of radiotherapy
  Acute toxicity according to CTCAE v. 4.0. This will record any reasons why balloon insertion is not possible for review.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Stratford, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital NHS Foundation Trust, Manchester, Manchester, United Kingdom